CLINICAL TRIAL: NCT05001074
Title: Randomized Controlled Trial Comparing Immediate Versus Extended Release Tacrolimus; Reducing Calcineurin Inhibitor Related Toxicity in Lung Transplantation Patients
Brief Title: Trial Comparing Immediate Versus Extended Release Tacrolimus; Reducing Calcineurin Inhibitor Related Toxicity in Lung Transplantation Patients
Acronym: REVOLUTION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heleen Grootjans (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor-Investigator, Heleen Grootjans, Drs. Heleen Grootjans, internist-nephrologist, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000134
Record Dates: First submitted 2021-07-01; First posted 2021-08-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Lung Transplant; Complications
Keywords: lung transplantation; chronic kidney disease; cardiovascular disease; extended release tacrolimus; LCP tacrolimus; immediate release tacrolimus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: De novo cohort, 2 arms: de novo lung transplant recipients. Conversion cohort, 2 arms: stable lung transplant recipients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- de novo cohort, extended release tacrolimus (Experimental): de novo cohort, extended release tacrolimus
  Interventions: Drug: Extended release tacrolimus
- de novo cohort, immediate release tacrolimus (Active Comparator): de novo cohort, immediate release tacrolimus
  Interventions: Drug: Immediate release tacrolimus
- conversion cohort, extended release tacrolimus (Experimental): conversion cohort, extended release tacrolimus
  Interventions: Drug: Extended release tacrolimus
- conversion cohort, immediate release tacrolimus (Active Comparator): conversion cohort, immediate release tacrolimus
  Interventions: Drug: Immediate release tacrolimus

INTERVENTIONS:
Drug: Extended release tacrolimus — de novo cohort: participants are randomised for extended release tacrolimus or immediate release tacrolimus direct post-lung transplantation Conversion cohort: participants are randomised for extended release tacrolimus or immediate release tacrolimus when >1 year post-lungtransplantation and with stable graft function
  Other Names: LCP tacrolimus
  Arms: conversion cohort, extended release tacrolimus; de novo cohort, extended release tacrolimus
Drug: Immediate release tacrolimus — de novo cohort: participants are randomised for extended release tacrolimus or immediate release tacrolimus direct post-lung transplantation Conversion cohort: participants are randomised for extended release tacrolimus or immediate release tacrolimus when >1 year post-lungtransplantation and with stable graft function
  Arms: conversion cohort, immediate release tacrolimus; de novo cohort, immediate release tacrolimus

SUMMARY:
Lung transplantation is a life-saving option in patients with end-stage lung disease. The introduction of calcineurin inhibitors has significantly improved long-term outcome in lung transplantation. The most frequently used calcineurin inhibitor as maintenance therapy is immediate release tacrolimus, dosed twice daily, which has shown to reduce both acute and chronic rejection. However, a drawback to the administration of tacrolimus is its toxicity. Especially progressive renal toxicity, new onset diabetes and hypertension contribute to the high cardiovascular burdon in this patient group. Since a few years an once daily extended release tacrolimus has been introduced in solid organ transplantation. The advantage of extended release tacrolimus is its prolonged release and higher bioavailability than other tacrolimus formulations. This result in lower peaks, more stable serum levels over 24 hours, and less fluctuation of blood concentrations.

Long-term toxicity outcome of extended release tacrolimus after lung transplantation has not been studied so far. Therefore the potential benefit of exteded release tacrolimus in de novo and stable post-lung transplant recipients should be investigated.

DETAILED DESCRIPTION:
Lung transplantation is a life-saving option in patients with end-stage lung disease. The introduction of calcineurin inhibitors (CNI) has significantly improved long-term outcome in lung transplantation. The most frequently used CNI as maintenance therapy is immediate release tacrolimus, dosed twice daily, which has shown to reduce both acute and chronic rejection. However, a drawback to the administration of tacrolimus is its toxicity. Especially progressive renal toxicity, new onset diabetes and hypertension contribute to the high cardiovascular burdon in this patient group. In lung transplant recipients the incidence of severe renal impairment, new onset of diabetes mellitus, hypertension and dyslipidemia is 53,9%, 40%, 80% and 40,3% post lung transplantation. Tremor is one of the most common CNI induced neurological toxic effect, besides polyneuropathy, headaches, insomnia, vertigo, dysesthesia and reduced cognitive ability. These complications are, among others, attributed to high peak serum tacrolimuslevels, whereas the effectiveness of the drug is determined by the area under the curve. In general lung transplant recipients have higher peak and trough levels when compared to other solid organ transplant recipients and therefore potentially experience more severe toxic side effects.

Since a few years an once daily extended release tacrolimus has been introduced in solid organ transplantation. The advantage of extended release tacrolimus is its prolonged release and higher bioavailability than other tacrolimus formulations. This result in lower peaks, more stable serum levels over 24 hours, and less fluctuation of blood concentrations. In addition, for an equal overall systemic tacrolimus exposure a 30% lower dosage is needed for extended release tacrolimus when compared to other formulations. In kidney and liver transplantation, extended release tacrolimus is safe and effective. Langone et al demonstrated in an enriched population of kidney transplant patients with tremor, that extended release tacrolimus improved hand tremor compared to immediate release tacrolimus.

Long-term toxicity outcome of extended release tacrolimus after lung transplantation has not been studied so far. Therefore the potential benefit of exteded release tacrolimus in de novo and stable post-lung transplant recipients should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Single or bilateral lung transplantation
* On twice daily tacrolimus with stable trough levels in target range
* Participant in the TransplantLines biobank study in the UMCG

Additional criteria for Conversion cohort:

* At least one year after lung transplantation with a stable clinical course and lung function
* eGFR >30ml/min*1.73m2 calculated with the CKD-EPI formula

Exclusion Criteria:

* Administration of mTOR inhibitors; everolimus, sirolimus
* Quadruple immunosuppression
* Renal transplantation
* The subject has any disease or condition that might interfere with completion of this study or reaching the primary endpoint (e.g., life expectancy of <3 years, renal replacement therapy at start study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
renal function: absolute change in eGFR | 2 years
  absolute change in eGFR absolute change in eGFR change in eGFR at 2 years

SECONDARY OUTCOMES:
graft function | 2 years
  Acute graft dysfunction is a clinical diagnoses, with or without histological confirmation, and indictation for rejection treatment such as methylprednisolon. Chronic graft dysfunction is defined according to the ISHLT guidelines, as a persistent decline (≥20%) in measured FEV1 value from baseline.
renal function: 40% eGFR reduction | 2 years
  40% eGFR reduction
renal function: 50% eGFR reduction | 2 years
  50% eGFR reduction
renal function:end stage kidney disease | 2 years
  end stage kidney disease
hypertension | 2 years
  Incidence of inadequate regulated or new onset of hypertension
diabetes mellitus | 2 years
  Incidence of inadequate glycemic control of preexisting diabetes mellitus or new onset diabetes after transplantation (NODAT)
Infections | 2 years
  Incidence of infections
Malignancies | 2 years
  Incidence of malignancies
neurological function: tremor | 2 years
  Incidence of or change in pre-existing hand tremor by using the validated Fahn-Tolosa-Martin (FTM) tremor rating scale (grades of tremor 0-4, in which 0 indicated no tremor and 4 severe tremor)
neurological function: polyneuropathy | 2 years
  Incidence of or change in pre-existing polyneuropathy
neurological function: sleep quality | 2 years
  Incidence of or change in sleep quality by using validated questionnaire: Pittsburg Sleep Quality Index (PSQI)
neurological function: cognitive functioning | 2 years
  Incidence of or change in cognitive functioning by using validated questionnaire: the Cognitive Functioning Questionnaire (CFQ)
quality of life score | 2 years
  change in SF36 score
pharmacogenetic | 2 years
  explorative endpoints: effects of well known variances in CYP3A4, CYP3A5 and ABCB1 transporter function on tacrolimus metabolism (resulting in so-called slow and fast tacrolimus metabolisers) on long-term tacrolimus renal toxicity by using absolute eGFR change
pharmacogenetic | 2 years
  explorative endpoints: effects of well known variances in CYP3A4, CYP3A5 and ABCB1 transporter function on tacrolimus metabolism (resulting in so-called slow and fast tacrolimus metabolisers) on long-term tacrolimus neurological toxicity: change in incidence of or change in pre-existing hand tremor by using the validated Fahn-Tolosa-Martin tremor rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Tji Gan, Principal Investigator — University Medical Center Groningen
Locations (1):
- University medical center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sintes H, Saez-Gimenez B, Berastegui C, Lopez-Meseguer M, Monforte V, Bravo C, Vima J, Gomez-Olles S, Roman A. Pharmacokinetic Study of Conversion Between 2 Formulations of Once-daily Extended-release Tacrolimus in Stable Lung Transplant Patients. Transplantation. 2018 Oct;102(10):e439-e446. doi: 10.1097/TP.0000000000002348. PMID 29965950
- [Result] Mendez A, Berastegui C, Lopez-Meseguer M, Monforte V, Bravo C, Blanco A, Camos S, Pou L, Roman A. Pharmacokinetic study of conversion from tacrolimus twice-daily to tacrolimus once-daily in stable lung transplantation. Transplantation. 2014 Feb 15;97(3):358-62. doi: 10.1097/01.TP.0000435699.69266.66. PMID 24492423
- [Result] TruneCka P, Klempnauer J, Bechstein WO, Pirenne J, Friman S, Zhao A, Isoniemi H, Rostaing L, Settmacher U, Monch C, Brown M, Undre N, Tisone G; DIAMONDdagger study group. Renal Function in De Novo Liver Transplant Recipients Receiving Different Prolonged-Release Tacrolimus Regimens-The DIAMOND Study. Am J Transplant. 2015 Jul;15(7):1843-54. doi: 10.1111/ajt.13182. Epub 2015 Feb 23. PMID 25707487
- [Result] Sanchez Fructuoso A, Ruiz JC, Franco A, Diekmann F, Redondo D, Calvino J, Serra N, Aladren MJ, Cigarran S, Manonelles A, Ramos A, Gomez G, Gonzalez Posada JM, Andres A, Beneyto I, Muniz AL, Perello M, Lauzurica R. Effectiveness and safety of the conversion to MeltDose(R) extended-release tacrolimus from other formulations of tacrolimus in stable kidney transplant patients: A retrospective study. Clin Transplant. 2020 Jan;34(1):e13767. doi: 10.1111/ctr.13767. Epub 2019 Dec 31. PMID 31815310